CLINICAL TRIAL: NCT04145895
Title: Postoperative Activity Restrictions in Children
Acronym: PARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Pavan Brahmamdam, Pediatric Surgeon, Corewell Health East
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-224
Record Dates: First submitted 2019-10-25; First posted 2019-10-31 (Actual); Results first posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-05

CONDITIONS: Pediatric Post-operative Time to Return to Full Activity
Keywords: Post-operative activity restriction; Pediatric inguinal hernia repair; Pediatric laparoscopic appendectomy

STUDY DESIGN:
Intervention Model Description: Prospective, nonrandomized, parallel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physician-directed Postoperative Activity Restriction (Other): Postoperative activity restrictions prescribed by physician.
  Interventions: Other: Postoperative activity restrictions
- Self-directed Postoperative Activity Restriction (Other): Postoperative activity restrictions self-determined (parent/guardian and/or patient).
  Interventions: Other: Postoperative activity restrictions

INTERVENTIONS:
Other: Postoperative activity restrictions — Recommendations for return to full activity including return to school, sports, exercise, etc.

SUMMARY:
This study will investigate the need for and length of postoperative activity restrictions in children following a laparoscopic appendectomy or inguinal hernia repair. Currently, no consensus exists and restrictions are based on doctors' experience and preference. Children and their parents/guardians will decide if they wish to participate in this study. Those who wish to participate and who are eligible to participate will decide which postoperative activity restrictions they would like the child to follow. The child will follow either 1) doctor-directed restrictions or 2) self-directed restrictions.A parent or guardian will complete a survey 1-3 months after the procedure, to assess patient and family satisfaction and patient outcome.

DETAILED DESCRIPTION:
Postoperative activity restrictions minimize the risk of surgical complications and prevent stress on the operative site. In the pediatric population, surgeons may restrict school attendance, participation in playground or gym, and participation in contact sports or heavy lifting. Currently, surgeons give pediatric patients postoperative restrictions following routine pediatric procedures (laparoscopic appendectomy and inguinal hernia repair) without evidence-based clinical practice guidelines. However, there is considerable variability amongst surgeons. It is common practice to provide some level of postoperative restrictions, which are primarily based on the surgeon's experience.While many surgeons prescribe specific postoperative instructions, some recommend self-directed restrictions. Self-directed restrictions instruct that the child return to school and normal physical activity when they and parents feel they are able to do so. There is no evidence that this practice is associated with any adverse outcomes.

This study will utilize a convenience sample of pediatric patients treated at Beaumont Royal Oak and Troy for routine inguinal hernia repair and laparoscopic appendectomy. There will be two populations: patients undergoing the procedures (Patient population) and their parents/guardians (Parent population) who will be completing the postoperative survey. Both parents/guardians and children were enrolled.

The Principal Investigator will review the operating room schedule and identify patients who are scheduled for either of the two procedures. Parents and patients who are eligible to participate in the study will be approached, the study explained and voluntary consent obtained. The participants will be provided an information sheet detailing the study, the risks, and the benefits. The researchers will describe the two groups the participant can enroll in. If the parents decide to enroll their child in the study they will then choose to be in either the control group (physician-directed) or the variable group (self-directed). The control group will be those individuals who choose physician-directed instructions which detail that they can resume all normal activity 2 weeks after their procedure. The experimental group will be those individuals who choose self-directed instructions which specify that they may return to full activity when their pain is improving and the parent feels comfortable with them doing so. For each group, the family will be provided with discharge instructions, a copy of these discharge instructions are provided in the study documents. A parent or guardian will complete a postoperative survey 1-3 months post procedure. The survey will assess: time of pain medication, time to return to school, time to resume full activity, wound healing, postoperative complications, changes in pain, compliance with instructions, patient satisfaction, time parent took off from work, if additional childcare was needed following the procedure, and parental satisfaction with the procedure and postoperative instructions.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Patient being treated at Royal Oak or Troy Beaumont for a routine inguinal hernia repair or appendectomy
* For inguinal hernia repair: 2-13 years of age
* For appendectomy: less than 18 years

Exclusion Criteria for Patients:

* Older than 18 years of age upon admission
* Patients with perforated or complicated appendicitis
* For laparoscopic appendectomy: patient required a conversion to open appendectomy
* Patient experienced a complicated procedure or concomitant operation

Inclusion Criteria for Parent/Guardians:

* 18 years or older
* Their child meets the inclusion criteria for participation in this study

Exclusion Criteria for Parent/Guardians:

* Less than 18 years of age
* Their child does not meet the inclusion criteria for participation in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavan Brahmamdam, MD, Principal Investigator — Corewell Health East
Locations (2):
- United States (2):
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital, Troy, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baumann LM, Williams K, Ghomrawi H, Abdullah F. Current practice patterns for postoperative activity restrictions in children. J Pediatr Surg. 2019 Jul;54(7):1432-1435. doi: 10.1016/j.jpedsurg.2018.06.025. Epub 2018 Jun 26. PMID 30146309

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total enrollment numbers represent both children and parents/guardians.
Period: Overall Study
Arm/Group | Physician-directed Postoperative Activity Restriction | Self-directed Postoperative Activity Restriction
Started | 42 | 126
Completed | 40 | 124
Not Completed | 2 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Ages were collected from children only. Baseline data was not collected for parents/guardians.
Groups:
- Total: Total of all reporting groups
Arm/Group | Physician-directed Postoperative Activity Restriction | Self-directed Postoperative Activity Restriction | Total
Number analyzed (Participants) | 20 | 62 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.0 (4.4) | 11.3 (3.2) | 10.5 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 25 | 33
  Male | 12 | 37 | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 62 | 82

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Outcomes - Clinical Complications
Description: Number of child participants who developed post op complications
Time Frame: six weeks post op
Population: data analyzed only for child participants
Measure: Count of Participants; unit: Participants
Arm/Group | Physician-directed Postoperative Activity Restriction | Self-directed Postoperative Activity Restriction
Number analyzed (Participants) | 20 | 62
Participants | 2 | 5

2. Primary Outcome: Post Operative Outcomes - Patient Satisfaction (Combination of Child, Parent and Satisfaction With Discharge Guidelines)
Description: Median satisfaction score ranging from 0-12 on a scale where 0=very satisfied, 1= satisfied, 2= neither satisfied nor dissatisfied, 3= dissatisfied, 4= very dissatisfied, and defined as combination of child + parent + discharge guidelines satisfaction ratings. Lower numbers = more satisfaction.
Time Frame: six weeks post op
Population: Both children and parents completed satisfaction surveys. Satisfaction data available only for the n=106 who completed the post-op survey.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Physician-directed Postoperative Activity Restriction | Self-directed Postoperative Activity Restriction
Number analyzed (Participants) | 22 | 84
score on a scale | 0 [0 to 1] | 0 [0 to 5]

3. Primary Outcome: Post Operative Outcomes - Length of Time to Return to Full Activity
Description: Mean/Standard deviation (SD) number of days to return to full activity
Time Frame: six weeks post op
Population: Data analyzed for child participants with survey responses.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Physician-directed Postoperative Activity Restriction | Self-directed Postoperative Activity Restriction
Number analyzed (Participants) | 11 | 41
days | 11.9 (7.5) | 8.9 (5.3)

4. Secondary Outcome: Number of Parents/Guardians Choosing Self-directed Post Operative Instructions
Description: Number of parents/guardians who chose self-directed post operative instructions
Time Frame: six weeks post op
Population: data analyzed only for parent/guardian participants
Measure: Count of Participants; unit: Participants
Arm/Group | Physician-directed Postoperative Activity Restriction | Self-directed Postoperative Activity Restriction
Number analyzed (Participants) | 20 | 62
Participants | 0 | 62

5. Secondary Outcome: Number of Parent/Guardians Choosing Physician-directed Post Operative Instructions
Description: Number of parent/guardian who chose physician-directed post operative instructions
Time Frame: six weeks post op
Population: data analyzed only for parent/guardian participants
Measure: Count of Participants; unit: Participants
Arm/Group | Physician-directed Postoperative Activity Restriction | Self-directed Postoperative Activity Restriction
Number analyzed (Participants) | 20 | 62
Participants | 20 | 0

6. Secondary Outcome: Number of Parental Days Off Work Taken in the Self-directed Post Operative Course Group Versus Physician-directed Course Group
Description: Mean/SD number of days parents took off work during the post operative period
Time Frame: six weeks post op
Population: data analyzed for parents who reported taking time off in survey
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Physician-directed Postoperative Activity Restriction | Self-directed Postoperative Activity Restriction
Number analyzed (Participants) | 10 | 36
days | 2.1 (4.3) | 1.4 (2.7)

ADVERSE EVENTS:
Time Frame: 6 months post procedure
Description: adverse event data not collected from parents
Arm/Group | Physician-directed Postoperative Activity Restriction | Self-directed Postoperative Activity Restriction
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/62
Other Adverse Events (participants affected / at risk) | 2/20 | 5/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physician-directed Postoperative Activity Restriction (N=20) | Self-directed Postoperative Activity Restriction (N=62)
infection requiring antibiotics (Infections and infestations) | 1 (1) | 2 (2)
anesthesia reaction (Surgical and medical procedures) | 1 (1) | 0 (0)
skin inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
drug rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/95/NCT04145895/Prot_SAP_000.pdf